CLINICAL TRIAL: NCT04983862
Title: Phase I Trial of Real-Time Intraoperative Fluorescent Imaging of Nerve Structures Using Illuminare-1, A Novel Myelin-Binding Fluorophore
Brief Title: Fluorescent Imaging of Nerves With Illuminare-1 During Surgery
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: Illuminare Biotechnologies (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 21-099
Record Dates: First submitted 2021-07-22; First posted 2021-07-30 (Actual); Last update posted 2025-09-16 (Actual); Status verified 2025-09

CONDITIONS: Prostate Adenocarcinoma
Keywords: Fluorescent Imaging; Illuminare-1; Myelin-Binding Fluorophore; 21-099

STUDY DESIGN:
Intervention Model Description: This is a first-in-human, single-arm, open-label, dose-escalation phase I study to investigate the safety of Illuminare-1, a myelin-binding fluorescent small molecule in patients undergoing routine minimally invasive radical prostatectomy.
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: Yes

ARMS (1):
- Illuminare-1 (Experimental)
  Interventions: Drug: Illuminare-1; Device: Karl Storz D-Light C photodynamic diagnostic (PDD)

INTERVENTIONS:
Drug: Illuminare-1 — Illuminare-1 at 3 dose levels in patients undergoing minimally invasive radical prostatectomy and bilateral pelvic lymph node dissection. Dose levels of the agent will be administered starting at 0.25mg/kg, with increases in dose between cohorts of no more than 0.75 mg/kg until a maximum dose of 3.0mg/kg is reached, if needed. At the dose identified to have the acceptable NMR and no associated DLTs, Illuminare-1 will be studied in up to 20 additional patients at this dose to optimize the imaging protocol and provide additional safety data.
Device: Karl Storz D-Light C photodynamic diagnostic (PDD) — The Storz PDD system will be used as the hardware system in this phase 1 study due to its proven safety profile.

SUMMARY:
This study will test the safety of using Illuminare-1 during standard surgery for prostate cancer. The study researchers will test increasing doses of Illuminare-1 to find the dose that makes the nerve structures fluoresce (light up) but causes few or mild side effects. When the researchers find this dose, it will be tested in new groups of study participants to see whether surgery performed using Illuminare-1 guidance is better than surgery performed without intraoperative guidance. The researchers will also do tests to study the way the body absorbs, distributes, and gets rid of Illuminare-1. This study is the first to test Illuminare-1 in people. Illuminare-1 has received Fast Track designation from the US FDA.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older and capable of signing their own consent form
* Scheduled for minimally invasive radical prostatectomy with pelvic lymph node dissection

Exclusion Criteria:

* Prior pelvic surgery or pelvic radiation therapy
* Known central nervous or peripheral nervous system disease or insult (including neurodegenerative diseases), current use of neurotoxic medications, or use of cytotoxic chemotherapy with known neurotoxicity within 1 month
* Exposure to investigational agents in the immediate 30 days before or 15 days after study drug administration
* Patients with significant renal dysfunction (<60 mL/min as assessed by the Cockcroft Gault calculation for creatinine clearance)
* Clinically significant hepatic/liver impairment (liver function tests more than 2x institutional normal upper limit)
* Exposure to phototoxic drugs such as St. John's wort, griseofulvin, thiazide diuretics, sulfonylureas, phenothiazines, sulphonamides, quinolones, and tetracyclines, should be avoided. If safe to discontinue use for a limited time, patients may participate on this trial but will discontinue the use of the interfering drug for 5 half-lives before Illuminare-1 injection to permit full washout, as well as for 48 hours after administration of Illuminare-1.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Prostate cancer
Enrollment: 41 (Actual)
Dates: Start 2021-10-04 (Actual); Primary Completion 2025-09-09 (Actual); Study Completion 2025-09-09 (Actual)

PRIMARY OUTCOMES:
determine the safety of Illuminare-1 | up to 45 days
  Five patients will be observed at each dose level. If > 20% of patients within a cohort experience a grade 2 or higher adverse event that is considered attributable to the drug and clinically significant, dose escalation will be stopped at that level, and the prior dose level will be considered the MTD. DLTs will be defined using NCI-CTCAE 5.0.

CONTACTS AND LOCATIONS:
Overall Officials: Timothy Donahue, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (6):
- United States (6):
  - Memorial Sloan Kettering Basking Ridge (Limited Protocol Activities), Basking Ridge, New Jersey
  - Memorial Sloan Kettering Monmouth (Limited protocol activities), Middletown, New Jersey
  - Memorial Sloan Kettering Bergen (Limited Protocol Activities), Montvale, New Jersey
  - Memorial Sloan Kettering Cancer Commack (Limited Protocol Activities), Commack, New York
  - Memorial Sloan Kettering Westchester (Limited protocol activities), Harrison, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York

IPD SHARING:
Plan to Share IPD: Yes
Memorial Sloan Kettering Cancer Center supports the international committee of medical journal editors (ICMJE) and the ethical obligation of responsible sharing of data from clinical trials. The protocol summary, a statistical summary, and informed consent form will be made available on clinicaltrials.gov when required as a condition of Federal awards, other agreements supporting the research and/or as otherwise required. Requests for deidentified individual participant data can be made beginning 12 months after publication and for up to 36 months post publication. Deidentified individual participant data reported in the manuscript will be shared under the terms of a Data Use Agreement and may only be used for approved proposals. Requests may be made to: crdatashare@mskcc.org.

REFERENCES:
- [Derived] Gold SA, Pere MM, Assel M, Doudt AD, Durdin TD, Silagy AW, Dean LW, Recabal P, Levine E, Burke A, Ragupathi G, Marzabadi MR, Yao ZK, Yang G, Yang G, Ouerfelli O, McCarter M, Chen X, Tzatha E, Coleman JA, Goh AC, Smith RC, Ehdaie B, Vickers AJ, Scardino PT, Eastham JA, Laudone VP, Donahue TF. Rizedisben in Minimally Invasive Surgery: A Nonrandomized Clinical Trial. JAMA Surg. 2025 Aug 1;160(8):875-883. doi: 10.1001/jamasurg.2025.1987. PMID 40601345
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org/mskcc/html/44.cfm